CLINICAL TRIAL: NCT00053794
Title: A Phase II Study Of Perifosine (D-21266) In Patients With Previously Untreated Metastatic Or Locally Advanced Soft Tissue Sarcoma
Brief Title: Perifosine in Treating Patients With Metastatic or Locally Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I155; CAN-NCIC-IND155 (Other: PDQ); CDR0000269476 (Other: PDQ)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Endometrial Cancer; Sarcoma
Keywords: adult alveolar soft-part sarcoma; adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult synovial sarcoma; endometrial stromal sarcoma; uterine leiomyosarcoma; adult malignant hemangiopericytoma; stage III adult soft tissue sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent adult soft tissue sarcoma; recurrent uterine sarcoma; adult malignant fibrous histiocytoma; adult neurofibrosarcoma; adult rhabdomyosarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Sarcoma; Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Sarcoma, Synovial; Sarcoma, Endometrial Stromal; Hemangiopericytoma, Malignant; Histiocytoma, Malignant Fibrous; Neurofibrosarcoma; Rhabdomyosarcoma | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perifosine in treating patients who have metastatic or locally advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of perifosine, in terms of response rate and duration of response, in patients with untreated metastatic or locally advanced soft tissue sarcoma.
* Determine the toxicity of this drug in these patients.
* Determine the early progression rate in patients treated with this drug.

OUTLINE: This is a non-randomized, non-blinded, multicenter study.

Patients receive a loading dose of oral perifosine twice on day 1 and then once daily on days 2-21 for the first course. For all subsequent courses, patients receive a loading dose of oral perifosine once on day 1 and then once daily on days 2-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for 1 month. Patients with stable or responsive disease are followed every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or locally advanced soft tissue sarcoma that is incurable by standard therapies, including any of the following types:

  * Uterine sarcomas

    * Mixed mesodermal
    * Leiomyosarcoma
    * Endometrial stromal sarcoma
  * Alveolar soft part sarcoma
  * Angiosarcoma/lymphangiosarcoma
  * Fibrosarcoma
  * Hemangiopericytoma
  * Leiomyosarcoma
  * Liposarcoma
  * Malignant fibrous histiocytoma
  * Neurogenic sarcoma
  * Pleomorphic rhabdomyosarcoma
  * Synovial sarcoma
  * Unclassifiable sarcoma
  * Undifferentiated sarcoma
* Excluded diseases include the following:

  * Bone sarcomas (e.g., osteosarcoma, Ewing's sarcoma, chondrosarcoma)
  * Embryonal rhabdomyosarcoma
  * Carcinosarcoma
  * Kaposi's sarcoma
  * Malignant mesothelioma
  * Neuroblastoma
  * Gastrointestinal stromal tumor
* At least 1 unidimensionally measurable site of disease (outside the previously irradiated area) defined as:

  * At least 20 mm by x-ray or physical exam
  * At least 10 mm by spiral CT scan
  * At least 20 mm by non-spiral CT scan NOTE: Bone lesions are not considered measurable

NOTE: Patients whose sole site of disease is within a previously irradiated area are allowed if there is evidence of progression or new lesions in the irradiated field

* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 2.5 times ULN

Renal

* Creatinine no greater than ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to perifosine
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No active or ongoing infection
* No psychiatric illness or social situation that would limit compliance with study requirements
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy for metastatic or locally advanced disease
* At least 6 months since prior adjuvant chemotherapy
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy (except low-dose, non-myelosuppressive radiotherapy)
* No concurrent radiotherapy to the sole site of measurable disease or for progressively symptomatic disease

Surgery

* At least 4 weeks since prior major surgery

Other

* No other concurrent anticancer therapy or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-06-09 (Actual); Primary Completion 2004-09-18 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Eisenhauer, MD, Study Chair — Cancer Centre of Southeastern Ontario at Kingston General Hospital
Locations (6):
- Canada (6):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knowling M, Blackstein M, Tozer R, Bramwell V, Dancey J, Dore N, Matthews S, Eisenhauer E. A phase II study of perifosine (D-21226) in patients with previously untreated metastatic or locally advanced soft tissue sarcoma: A National Cancer Institute of Canada Clinical Trials Group trial. Invest New Drugs. 2006 Sep;24(5):435-9. doi: 10.1007/s10637-006-6406-7. PMID 16528479